CLINICAL TRIAL: NCT05939505
Title: The Effect of Sujok Therapy on Symptom Burden and Comfort Level in Patients Undergoing Hemodialysis Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Candan DOGAN (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Sponsor-Investigator, Candan DOGAN, Instructor, Tokat Gaziosmanpasa University
Organization: Tokat Gaziosmanpasa University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: GaziosmanpasaU-HMŞRLK-CD-01
Record Dates: First submitted 2023-06-15; First posted 2023-07-11 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Dialysis; Complications
Keywords: dialysis, Su Jok therapy, nursing

STUDY DESIGN:
Intervention Model Description: randomized-controlled,placebo
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not know which group they are in. The person who analyzes the data obtained at the end of the study will not know the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Su Jok Therapy Group (Experimental): Su jok Therapy According to Sujok therapy, sujok therapy will be applied 14 times with an interval of one day with Mexican bean seeds on the points representing the kidney.
  Interventions: Other: Su Jok therapy; Other: routine interventions
- placebo group (Placebo Comparator): Instead of the Mexican bean seed used in Sujok therapy, plastic beans will be applied 14 times with an interval of one day.
  Interventions: Other: placebo; Other: routine interventions
- Control group (Active Comparator): Routine applications will be made in the Dialysis Unit.
  Interventions: Other: routine interventions

INTERVENTIONS:
Other: Su Jok therapy — Sujok therapy will be applied with Mexican bean seeds 14 times with an interval of one day.
  Arms: Su Jok Therapy Group
Other: placebo — Instead of the Mexican bean seed applied in sujok therapy, plastic beans will be applied 14 times with an interval of one day.
  Arms: placebo group
Other: routine interventions — routine applications in the hemodialysis unit

SUMMARY:
Many symptoms such as fatigue, muscle cramps, dry mouth, and headache that develop in patients due to the hemodialysis treatment process affect the quality of life and comfort of people. Sujok therapy is an effective method in symptom management. Although sujok therapy is an uncomplicated acupressure, it has positive features such as being uncomplicated so that it can be applied by the patients themselves.

This study is planned as a single-blind placebo-controlled randomized trial. Research Hypotheses H0/1: Hydrotherapy has no effect on symptom burden in hemodialysis patients. H0/2: Hydrotherapy has no effect on hemodialysis comfort in hemodialysis patients.

H1/1: Hydrotherapy has an effect on symptom burden in hemodialysis patients. H1/2: Hydrotherapy has an effect on hemodialysis comfort in hemodialysis patients.

Inclusion criteria of volunteers

1. 18 years or older
2. To be on HD treatment for at least 6 months In our study, there are three groups as experimental, placebo and control groups.

Group application steps to be applied water jok therapy(experimental groups); The right foot in men and the left foot in women will be preferred, and the outer and inner surface of the foot will be massaged with a massage stick for an average of 3 minutes, then the middle of the area between the 3rd and 4th toes and the wrist line on the outer surface of the foot, which represents the kidney area in the macro system. The pain point will be determined with a diagnostic metal rod in the thoracic 12th spine and the area representing the lumbar 3rd spine region, and it will be fixed with the help of a Mexican bean seed patch in the appropriate size for the painful spot, and it will be ensured to remain in the area for at least 8 hours.

Group administration steps to be administered placebo ( Placebo Groups); It is planned that all the application steps will be the same as the group in which water jok therapy was applied, but instead of Mexican bean seeds, the use of red plastic number bean, which is used to improve the counting skill, is planned.

Control group application steps; It is planned to implement routine interventions applied in dialysis centers.

Sujok therapy and placebo application will be applied by the researcher during each dialysis session and it is planned to be carried out in a way to complete 14 sessions.

In the study, it is planned to use Dialysis Symptom Index together with Hemodialysis Comfort Scale Version Ⅱ for the groups before the application, after the seventh and fourteenth application.

DETAILED DESCRIPTION:
The purpose of hemodialysis treatment; to remove metabolic wastes from the blood, to reduce symptoms and complications in patients, and to increase life expectancy and quality. During the hemodialysis treatment process, many comorbidities, complications and symptoms may occur in patients(1). The number of symptoms and the high load of effects in patients negatively affect their quality of life. In addition, life expectancy decreases and mortality rates increase in these patients (2). In order to reduce the burden of symptoms accompanying HD and increase the quality of life, it is necessary to ensure HD sufficiency and maintain physical, mental and biochemical well-being Su Jok therapy is defined as a modern interpretation of acupressure/acupuncture that can be applied to both acute and chronic diseases for symptom improvement and health promotion by using reflection points on the hands and feet(3). According to the Su Jok theory; There is energy flow and circulation in the body, and in case of illness, this energy flow is disrupted in the organ or a part of the body. With Su Jok therapy, it is argued that as a result of the application of various applicators (rings, metal starlets, magnets, etc.) and appropriate plant seeds to the hands and feet, which the energy system considers as stimulating points, the physically sick organ or body area is stimulated. It is stated that as a result of this stimulation, the energy in the body is activated and an improvement in symptoms is observed (4). Su Jok therapy, with the absence of any interference to the body, ease of application and learning, allows patients to apply it on their own with good counseling, and symptom management is also very effective. It is stated that nurses can apply Su Jok therapy as an integrative method in symptom management due to the simple and uncomplicated nature of Su Jok therapy and the need for invasive procedures (5).

Details of Study Design and Method This study is planned as a single-blind placebo-controlled randomized trial. The number of samples to be reached with patients who meet the criteria for inclusion in the study is planned to be the group in which sujok therapy was applied (37 people), the group that was administered placebo (37 people) and the control group (37 people) in which routine applications were made.

The researcher attended the Sujok Therapy Training given by the International Sujok Association between 08-28.11.2022. The content of the training consists of theoretical and practical information including the history of Su Jok, its mechanism of action, areas of use, basic information about Su Jok points.

Group application steps to be applied water jok therapy; The right foot in men and the left foot in women will be preferred, and the outer and inner surface of the foot will be massaged with a massage stick for an average of 3 minutes, then the middle of the area between the 3rd and 4th toes and the wrist line on the outer surface of the foot, which represents the kidney area in the macro system. The pain point will be determined with a diagnostic metal rod in the thoracic 12th spine and the area representing the lumbar 3rd spine region, and it will be fixed with the help of a Mexican bean seed patch in the appropriate size for the painful spot, and it will be ensured to remain in the area for at least 8 hours. It also plans insect (micro system) work simultaneously with the macro system, and the pain point is detected with a diagnostic metal rod in the lower 2/3 part of the 3rd node (the area representing the kidney region in the insect system) on the outer surface of the toes, and the appropriate size for the painful point is located in Mexico. bean seed will be fixed with the help of a plaster and it will be ensured that it remains in the area for at least 8 hours.

Group administration steps to be administered placebo; It is planned that all the application steps will be the same as the group in which water jok therapy was applied, but instead of Mexican bean seeds, the use of red plastic number bean, which is used to improve the counting skill, is planned.

The right foot in men and the left foot in women will be preferred, and the outer and inner surface of the foot will be massaged with a massage stick for an average of 3 minutes, then the 3rd and 4th feet will be applied on the outer surface of the foot, which represents the kidney region in the macro system.

In the middle part of the area between the fingers and the wrist line (the area representing the thoracic 12th spine and the lumbar 3rd spine region), the pain point is detected with a diagnostic metal stick, and a plastic red counting bean in size suitable for the painful spot is fixed with the help of a plaster. It will be ensured to stay in the area for 8 hours. It also plans insect (micro system) work simultaneously with the macro system, and the pain point is detected with a diagnostic metal rod in the lower 2/3 of the 3rd knuckle (the area representing the kidney region in the insect system) on the outer surface of the toes, and plastic of the appropriate size for the painful point is determined. The red counting bean will be detected with the help of a plaster and it will be ensured to stay in the area for at least 8 hours.

Painful spot detection does not change until it is detected in the first session and the procedure is completed.

Control group application steps; It is planned to implement routine interventions applied in dialysis centers.

Sujok therapy and placebo application will be applied by the researcher during each dialysis session and it is planned to be carried out in a way to complete 14 sessions.

In the study, it is planned to use Dialysis Symptom Index together with Hemodialysis Comfort Scale Version Ⅱ for the groups before the application, after the seventh and fourteenth application.

Randomization Method Since the practitioner and the researcher evaluating the data are the same person in this study, double-blind approach cannot be used. Randomization will be done via https://www.randomizer.org/.

Data Collection Tools In collecting the data of the research;

* Personal Information Form prepared by the researcher, containing the socio-demographic characteristics of the patients,
* With Hemodialysis Comfort Scale Version Ⅱ
* Dialysis Symptom Index will be used.

Personal Information Form The personal information form prepared by the researchers is a form that includes the socio-demographic variables of the patients (age, gender, marital status), duration of hemodialysis treatment, and chronic disease status.

Hemodialysis Comfort Scale Version-II Since the hemodialysis comfort scale, which was first developed by Orak et al. in 2017, was insufficient, the scale was developed by Koşar Şahin and his friend in 2019, and the Hemodialysis Comfort Scale-Version II scale was created. The scale is a 5-point Likert-type scale consisting of 26 items and six sub-dimensions(6,7).

Dialysis Symptom Index Developed by Weisbord et al. in 2004, this scale assesses physical and emotional symptoms and their severity. The Turkish validity and reliability of the scale was done by the Foreword, Usta Yeşilbalkan(8,9) .

Data Collection The pre-test data of the study were planned to be collected during July 2023, after a brief information about the study was given to the individuals receiving dialysis treatment by the researcher. Pre-test data will be collected by the researcher by face-to-face interview method. Application of data collection forms takes an average of 25 minutes. "Personal Information Form", "Hemodialysis Comfort Scale Version-II," "Dialysis Symptom Index" will be applied to individuals in the control and experimental groups to collect data.

Collection of Post-Test Data:

Patients in the experimental group will be given a total of 14 sessions of water jok, 3 times a week for 5 weeks. Post-test data will be collected by applying Dialysis Symptom Index together with Hemodialysis Comfort Scale Version Ⅱ after the 7th and 14th sessions.

Patients in the placebo group will be given a total of 14 sessions of water jok, 3 times a week for 5 weeks. Post-test data will be collected by applying Dialysis Symptom Index together with Hemodialysis Comfort Scale Version Ⅱ after the 7th and 14th sessions.

From the collection of pre-test data on patients in the control group who did not undergo any intervention. After the 7th and 14th Sessions, posttest data will be collected by applying the Dialysis Symptom Index together with the Hemodialysis Comfort Scale Version Ⅱ to the patients.

ELIGIBILITY:
Inclusion Criteria:

* be 18 years or older
* Receiving hemodialysis treatment for at least 6 months
* agreeing to participate in the study

Exclusion Criteria:

* Having food, metal and plastic allergies
* Having a cognitive and psychiatric diagnosis
* Loss of sensation and amputation that prevents application in the feet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Symptom burden in hemodialysis patients | pre-therapy, up to 3 weeks, up to 5 weeks
  Dialysis Symptom Index

SECONDARY OUTCOMES:
hemodialysis comfort in hemodialysis patients | pre-therapy, up to 3 weeks, up to 5 weeks
  Hemodialysis Comfort Scale

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR